CLINICAL TRIAL: NCT00065468
Title: A Phase 3, Three-Arm, Randomized, Open-Label Study Of Interferon Alfa Alone, CCI-779 Alone, And The Combination Of Interferon Alfa And CCI-779 In First-Line Poor-Prognosis Subjects With Advanced Renal Cell Carcinoma.
Brief Title: Study Evaluating Interferon And CCI-779 In Advanced Renal Cell Carcinoma
Acronym: ARCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3066K1-304; NCT00070330 (obsolete NCT alias)
Record Dates: First submitted 2003-07-24; First posted 2003-07-25 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-09

CONDITIONS: Carcinoma, Renal Cell; Kidney Neoplasms
Keywords: Advanced Renal Cell Carcinoma; Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Interferon-alpha; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator)
  Interventions: Drug: Interferon Alfa
- B (Experimental)
  Interventions: Drug: CCI-779
- C (Experimental)
  Interventions: Drug: Interferon Alfa and CCI-779

INTERVENTIONS:
Drug: Interferon Alfa — Interferon alfa (Roferon) 3 MU given Sub Cutaneously three time /week for the first week, 9 MU given Sub Cutaneously three time /week for the second week, 18 MU given Sub Cutaneously three time /week thereafter.
  Arms: A
Drug: CCI-779 — 25 mg of CCI-779 given Intra Venously once per week
  Arms: B
Drug: Interferon Alfa and CCI-779 — 15 mg of CCI-779 given Intra Venously once per week; 6 MU of IFN alfa (Roferon) given Sub Cutaneously three time /week
  Arms: C

SUMMARY:
The primary objective of this study is efficacy. The primary efficacy endpoint of this study is a comparison of the overall survival of subjects treated with CCI-779 [Temsirolimus], administered intravenously [IV] once weekly and the combination of CCI-779, administered IV once weekly with Interferon Alfa [IFN alfa] subcutaneously [SC] three times per week [TIW], compared with the overall survival of subjects treated with IFN alfa (SC TIW) alone, in poor-prognosis subjects with advanced RCC.

ELIGIBILITY:
Inclusion Criteria:

* This study will be conducted in subjects with histologically confirmed, advanced (stage IV or recurrent disease) RCC who have not received prior systemic therapy for their disease,

Exclusion Criteria:

* Subjects with central nervous system (CNS) metastases
* Prior anticancer therapy for RCC
* Prior investigational therapy/agents within 4 weeks of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2003-07; Primary Completion 2006-06 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (141):
- United States (47):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, La Verne, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Urbana, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, South Bend, Indiana
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Great Falls, Montana
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, East Orange, New Jersey
  - Pfizer Investigational Site, Morristown, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Valhalla, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Seattle, Washington
- Argentina (6):
  - Pfizer Investigational Site, Buenos, Aires
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires
  - Pfizer Investigational Site, Córdoba, Córdoba Province
  - Pfizer Investigational Site, San Miguel de Tucumán, Tucumán Province
  - Pfizer Investigational Site, Mendoza
  - Pfizer Investigational Site, Quilmes
- Australia (7):
  - Pfizer Investigational Site, Kogarah, New South Wales
  - Pfizer Investigational Site, Newcastle, New South Wales
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Footscray, Victoria
  - Pfizer Investigational Site, Heidelberg, Victoria
  - Pfizer Investigational Site, Melbourne, Victoria
- Canada (14):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Newmarket, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Greenfield Park, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Hamilton, Ontario
- Czechia (2):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Prague
- Germany (3):
  - Pfizer Investigational Site, Bonn, North Rhine-Westphalia
  - Pfizer Investigational Site, Essen, North Rhine-Westphalia
  - Pfizer Investigational Site, Mainz, Rhineland-Palatinate
- Greece (2):
  - Pfizer Investigational Site, Heraklion, Creete
  - Pfizer Investigational Site, Pátrai
- Pfizer Investigational Site, Budapest, Hungary
- Italy (3):
  - Pfizer Investigational Site, Roma, RM
  - Pfizer Investigational Site, Foggia
  - Pfizer Investigational Site, Milan
- Latvia (2):
  - Pfizer Investigational Site, Daugavpils
  - Pfizer Investigational Site, Riga
- Pfizer Investigational Site, Vilnius, Lithuania
- Mexico (2):
  - Pfizer Investigational Site, Monterrey, Nuevo León
  - Pfizer Investigational Site, León
- Netherlands (3):
  - Pfizer Investigational Site, Nijmegen, GA
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Enschede
- Poland (8):
  - Pfizer Investigational Site, Bytom
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Olsztyn
  - Pfizer Investigational Site, Opole
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Siedlce
  - Pfizer Investigational Site, Warsaw
- Russia (6):
  - Pfizer Investigational Site, Barnaul
  - Pfizer Investigational Site, Kemerovo
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Obninsk
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Ufa
- Pfizer Investigational Site, Sremska Kamenica, Novi Sad, Serbia and Montenegro
- Pfizer Investigational Site, Belgrade, Serbia
- Slovakia (4):
  - Pfizer Investigational Site, Banská Bystrica
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Martin
  - Pfizer Investigational Site, Zlina
- South Africa (4):
  - Pfizer Investigational Site, Port Elizabeth, Eastern Cape
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Gauteng
- Spain (4):
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Oviedo, Principality of Asturias
- Sweden (3):
  - Pfizer Investigational Site, Stockholm, Sweden
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Uppsala
- Taiwan (4):
  - Pfizer Investigational Site, Taipei, ROC
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
  - Pfizer Investigational Site, Taoyuan District
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir
- Ukraine (6):
  - Pfizer Investigational Site, Dnietropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kiev
  - Pfizer Investigational Site, Lviv
  - Pfizer Investigational Site, Zaporizhzhya
- United Kingdom (4):
  - Pfizer Investigational Site, Manchester, Lancashire
  - Pfizer Investigational Site, Glasgow, Strathclyde
  - Pfizer Investigational Site, Sutton, Surrey
  - Pfizer Investigational Site, Nottingham
- Pfizer Investigational Site

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] de Velasco G, McKay RR, Lin X, Moreira RB, Simantov R, Choueiri TK. Comprehensive Analysis of Survival Outcomes in Non-Clear Cell Renal Cell Carcinoma Patients Treated in Clinical Trials. Clin Genitourin Cancer. 2017 Dec;15(6):652-660.e1. doi: 10.1016/j.clgc.2017.03.004. Epub 2017 Mar 21. PMID 28410911
- [Derived] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Derived] Grunwald V, McKay RR, Krajewski KM, Kalanovic D, Lin X, Perkins JJ, Simantov R, Choueiri TK. Depth of remission is a prognostic factor for survival in patients with metastatic renal cell carcinoma. Eur Urol. 2015 May;67(5):952-8. doi: 10.1016/j.eururo.2014.12.036. Epub 2015 Jan 7. PMID 25577718
- [Derived] Hudes G, Carducci M, Tomczak P, Dutcher J, Figlin R, Kapoor A, Staroslawska E, Sosman J, McDermott D, Bodrogi I, Kovacevic Z, Lesovoy V, Schmidt-Wolf IG, Barbarash O, Gokmen E, O'Toole T, Lustgarten S, Moore L, Motzer RJ; Global ARCC Trial. Temsirolimus, interferon alfa, or both for advanced renal-cell carcinoma. N Engl J Med. 2007 May 31;356(22):2271-81. doi: 10.1056/NEJMoa066838. PMID 17538086
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3066K1-304&StudyName=Study%20Evaluating%20Interferon%20And%20CCI-779%20In%20Advanced%20Renal%20Cell%20Carcinoma

RESULTS

PARTICIPANT FLOW:
Groups:
- Interferon Alfa: Interferon Alfa (Roferon) 3 million units (MU) subcutaneously 3 times per week for 1 week, then 9 MU subcutaneously 3 times per week for 1 week, then 18 MU subcutaneously 3 times per week until disease progression or treatment withdrawal
- Temsirolimus: Temsirolimus (CCI-779) 25 milligrams (mg) intravenously (IV) once per week until disease progression or treatment withdrawal
- Interferon Alfa and Temsirolimus: Interferon Alfa (Roferon) 6 MU subcutaneously 3 times per week and Temsirolimus (CCI-779) 15 mg IV once per week until disease progression or treatment withdrawal
Period: Overall Study
Arm/Group | Interferon Alfa | Temsirolimus | Interferon Alfa and Temsirolimus
Started | 207 | 209 | 210
Received Treatment | 200 | 208 | 208
Completed | 0 | 0 | 0
Not Completed | 207 | 209 | 210
Not completed — Death | 172 | 169 | 171
Not completed — Withdrawal by Subject | 3 | 4 | 5
Not completed — Lost to Follow-up | 5 | 3 | 2
Not completed — Discontinuation of study by Sponsor | 13 | 9 | 13
Not completed — Disease progression | 0 | 0 | 1
Not completed — Other | 14 | 24 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interferon Alfa | Temsirolimus | Interferon Alfa and Temsirolimus | Total
Number analyzed (Participants) | 207 | 209 | 210 | 626
Age Continuous [Mean (Standard Deviation); unit: years] | 59.2 (10.4) | 58.7 (10.0) | 59.3 (9.8) | 59.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 70 | 65 | 194
  Male | 148 | 139 | 145 | 432

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is the duration from randomization to death. For participants who are alive, overall survival is censored at the last contact.
Time Frame: Baseline up to Month 80
Population: Intent-to-treat (ITT) Population: all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Interferon Alfa | Temsirolimus | Interferon Alfa and Temsirolimus
Number analyzed (Participants) | 207 | 209 | 210
months | 7.3 [6.1 to 8.8] | 10.9 [8.6 to 12.7] | 8.4 [6.6 to 10.3]
Statistical Analysis 1: Comparison: Interferon Alfa vs Temsirolimus; Test type: Non-Inferiority or Equivalence — 2 null hypotheses (Ho) were tested: 1) Survival distributions for temsirolimus alone and Interferon Alfa (IFN)-alone treatment groups were identical. 2) Survival distributions for temsirolimus in combination with IFN and IFN-alone treatment groups were identical. The alternative hypothesis (Ha) for each test was that the survival distributions differed; p = 0.0252, Log Rank; Stratified by prior nephrectomy and region; Cox Proportional Hazard = 0.78, 95% CI 2-sided [0.63 to 0.97]
Statistical Analysis 2: Comparison: Interferon Alfa vs Interferon Alfa and Temsirolimus; Test type: Non-Inferiority or Equivalence — 2 null hypotheses (Ho) were tested: 1) Survival distributions for temsirolimus alone and IFN-alone treatment groups were identical. 2) Survival distributions for temsirolimus in combination with IFN and IFN-alone treatment groups were identical. The alternative hypothesis (Ha) for each test was that the survival distributions differed; p = 0.4902, Log Rank; Stratified by prior nephrectomy and region; Cox Proportional Hazard = 0.93, 95% CI 2-sided [0.75 to 1.15]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS based on Independent Central Review Assessment. The period from randomization until disease progression, death or date of last contact.
Time Frame: Baseline, monthly until tumor progression or death (up to Month 80)
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Interferon Alfa | Temsirolimus | Interferon Alfa and Temsirolimus
Number analyzed (Participants) | 207 | 209 | 210
months | 3.2 [2.2 to 4.0] | 5.6 [3.9 to 7.2] | 4.9 [3.9 to 6.0]
Statistical Analysis 1: Comparison: Interferon Alfa vs Temsirolimus; Test type: Superiority or Other; p = 0.0042, Log Rank; Stratified by prior nephrectomy and region; Cox Proportional Hazard = 0.74, 95% CI 2-sided [0.60 to 0.91]
Statistical Analysis 2: Comparison: Interferon Alfa vs Interferon Alfa and Temsirolimus; Test type: Superiority or Other; p = 0.0107, Log Rank; Stratified by prior nephrectomy and region; Cox Proportional Hazard = 0.76, 95% CI 2-sided [0.62 to 0.94]

3. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was the disappearance of all target lesions and non target lesions. PR was at least a 30 percent (%) decrease in sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Baseline, every 2 months until tumor progression or death (up to Month 80)
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interferon Alfa | Temsirolimus | Interferon Alfa and Temsirolimus
Number analyzed (Participants) | 207 | 209 | 210
percentage of participants | 5.3 [2.3 to 8.4] | 9.1 [5.2 to 13.0] | 9.5 [5.6 to 13.5]
Statistical Analysis 1: Comparison: Interferon Alfa vs Temsirolimus; Test type: Superiority or Other; p = 0.1361, Cochran-Mantel-Haenszel; Stratified by prior nephrectomy and region
Statistical Analysis 2: Comparison: Interferon Alfa vs Interferon Alfa and Temsirolimus; Test type: Superiority or Other; p = 0.1062, Cochran-Mantel-Haenszel; Stratified by prior nephrectomy and region

4. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical benefit: confirmed CR or PR or had stable disease (SD) lasting at least 24 weeks. CR was the disappearance of all target lesions and non target lesions. PR was at least a 30% decrease in sum of the LD of target lesions, taking as reference the baseline sum LD. SD was having neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Baseline, every 2 months until tumor progression or death (up to Month 80)
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interferon Alfa | Temsirolimus | Interferon Alfa and Temsirolimus
Number analyzed (Participants) | 207 | 209 | 210
percentage of participants | 16.4 [11.4 to 21.5] | 34.0 [27.6 to 40.4] | 30.0 [23.8 to 36.2]
Statistical Analysis 1: Comparison: Interferon Alfa vs Temsirolimus; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by prior nephrectomy and region
Statistical Analysis 2: Comparison: Interferon Alfa vs Interferon Alfa and Temsirolimus; Test type: Superiority or Other; p = 0.0011, Cochran-Mantel-Haenszel; Stratified by prior nephrectomy and region

5. Secondary Outcome: Duration of Response (DR)
Description: DR: Time from first documentation of objective tumor response to first date that recurrence or progressive disease (PD) was objectively documented, taking as a reference for PD, the smallest sum LD recorded since randomization.
Time Frame: Baseline, every month until tumor progression or death (up to Month 80)
Population: ITT subset of participants who had a response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Interferon Alfa | Temsirolimus | Interferon Alfa and Temsirolimus
Number analyzed (Participants) | 11 | 19 | 20
months | 7.4 [5.1 to 18.4] | 11.1 [9.1 to 13.8] | 9.3 [5.8 to 23.1]

6. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is defined as the time from the date of randomization to the date of PD or death, withdrawal from treatment due to an adverse event (AE), withdrawal of voluntary consent, or lost to follow-up, whichever occurred first, censored at the date of the conclusion of treatment phase.
Time Frame: Baseline, every month until tumor progression or death (up to Month 80)
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Interferon Alfa | Temsirolimus | Interferon Alfa and Temsirolimus
Number analyzed (Participants) | 207 | 209 | 210
months | 1.9 [1.7 to 1.9] | 3.7 [3.4 to 3.9] | 2.5 [1.9 to 3.6]
Statistical Analysis 1: Comparison: Interferon Alfa vs Temsirolimus; Test type: Superiority or Other; p < 0.0001, Log Rank; Stratified by prior nephrectomy and region; Cox Proportional Hazard = 0.62, 95% CI 2-sided [0.51 to 0.76]
Statistical Analysis 2: Comparison: Interferon Alfa vs Interferon Alfa and Temsirolimus; Test type: Superiority or Other; p = 0.0020, Log Rank; Stratified by prior nephrectomy and region; Cox Proportional Hazard = 0.73, 95% CI 2-sided [0.60 to 0.89]

7. Secondary Outcome: Quality-adjusted Time Without Symptoms or Toxicity (Q-TWiST)
Description: The Q-Twist is not a score calculated for each participant but is defined only on a by treatment group basis. For each treatment group, it is the weighted sum of the mean durations of the health states Tox, Twist, and Relapse. Tox is defined as time with severe toxicity related to treatment; Twist: time without symptoms or toxic side effects; and Relapse: time after relapse/progression. The mean duration of each health state is calculated based on the area under the Kaplan Meier curve pertaining to that health state. There is no direct method for calculating the "dispersion" of Q-Twist, and it is typically done using bootstrap method for purposes of inference (see, e.g., Glasziou PP, Simes RJ, Gelber RD. Quality adjusted survival analysis. Stat Med 1990; 9: 1259-76). In practice, as apparently in the case with this study, the intermediate values resulting from the bootstrap exercise were not displayed.
Time Frame: Baseline to Month 80
Population: ITT
Measure: Number; unit: months
Arm/Group | Interferon Alfa | Temsirolimus | Interferon Alfa and Temsirolimus
Number analyzed (Participants) | 207 | 209 | 210
months | 6.9083 | 8.3707 | 7.4821

8. Secondary Outcome: European Quality of Life Health Questionnaire (EQ-5D) - Index Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. EQ-5D index measured 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Range of EQ-5D index score = -0.594 to 1 where higher scores indicated a better health state.
Time Frame: Baseline
Population: ITT;(N)=participants with evaluable data. Week 12 and 32 data collected for individual participants but not summarized.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Interferon Alfa | Temsirolimus | Interferon Alfa and Temsirolimus
Number analyzed (Participants) | 197 | 204 | 197
units on a scale | 0.656 [-0.319 to 1.000] | 0.689 [-0.181 to 1.000] | 0.689 [-0.239 to 1.000]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a Serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another subject, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Interferon Alfa | Temsirolimus | Interferon Alfa and Temsirolimus
Serious Adverse Events (participants affected / at risk) | 99/200 | 82/208 | 122/208
Other Adverse Events (participants affected / at risk) | 197/200 | 208/208 | 205/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Alfa (N=200) | Temsirolimus (N=208) | Interferon Alfa and Temsirolimus (N=208)
ABDOMINAL PAIN (General disorders) | 1 | 5 | 4 — Body as a whole
BACK PAIN (General disorders) | 2 | 4 | 1
CARCINOMA (General disorders) | 9 | 4 | 13
ASTHENIA (General disorders) | 7 | 3 | 10
FEVER (General disorders) | 3 | 3 | 8
ASCITES (General disorders) | 1 | 2 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 2 | 1
PAIN (General disorders) | 0 | 2 | 3
ABSCESS (General disorders) | 1 | 1 | 0
ACCIDENTAL INJURY (General disorders) | 0 | 1 | 3
CHEST PAIN (General disorders) | 1 | 1 | 1
HERNIA (General disorders) | 0 | 1 | 0
INFECTION (General disorders) | 1 | 1 | 1
INFLAMMATION (General disorders) | 0 | 1 | 0
MALAISE (General disorders) | 1 | 1 | 0
MEDICATION ERROR (General disorders) | 0 | 1 | 0
NEOPLASM (General disorders) | 0 | 1 | 0
OVERDOSE (General disorders) | 0 | 1 | 2
PELVIC PAIN (General disorders) | 0 | 1 | 0
SEPSIS (General disorders) | 0 | 1 | 3
ABDOMINAL SYNDROME ACUTE (General disorders) | 0 | 0 | 1
ACCIDENTAL OVERDOSE (General disorders) | 0 | 0 | 1
ALLERGIC REACTION (General disorders) | 1 | 0 | 1
CELLULITIS (General disorders) | 1 | 0 | 3
CHILLS (General disorders) | 1 | 0 | 0
FLU SYNDROME (General disorders) | 0 | 0 | 1
GENERALIZED EDEMA (General disorders) | 1 | 0 | 0
NECK PAIN (General disorders) | 0 | 0 | 2
TUMOR LYSIS SYNDROME (General disorders) | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 2 | 1 — Cardiovascular system
CONGESTIVE HEART FAILURE (Cardiac disorders) | 1 | 2 | 0
DEEP VEIN THROMBOSIS (Cardiac disorders) | 1 | 2 | 0
HYPERTENSION (Cardiac disorders) | 1 | 2 | 2
MYOCARDIAL INFARCT (Cardiac disorders) | 2 | 2 | 1
PULMONARY EMBOLUS (Cardiac disorders) | 1 | 2 | 3
CEREBROVASCULAR ACCIDENT (Cardiac disorders) | 0 | 1 | 1
HEART FAILURE (Cardiac disorders) | 1 | 1 | 2
INTRACRANIAL HEMORRHAGE 0 (Cardiac disorders) | 0 | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 1 | 0
PERIPHERAL GANGRENE (Cardiac disorders) | 0 | 1 | 0
SYNCOPE (Cardiac disorders) | 0 | 1 | 0
TACHYCARDIA SINUS (Cardiac disorders) | 0 | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 1
CARDIOMYOPATHY (Cardiac disorders) | 0 | 0 | 1
CEREBRAL HEMORRHAGE (Cardiac disorders) | 0 | 0 | 1
CEREBRAL ISCHEMIA (Cardiac disorders) | 0 | 0 | 1
CEREBROVASCULAR DISORDER (Cardiac disorders) | 1 | 0 | 0
HEART ARREST (Cardiac disorders) | 0 | 0 | 1
HEMORRHAGE (Cardiac disorders) | 1 | 0 | 2
HYPOTENSION (Cardiac disorders) | 2 | 0 | 2
HYPOVOLEMIA (Cardiac disorders) | 1 | 0 | 0
POSTURAL HYPOTENSION 1 (Cardiac disorders) | 1 | 0 | 0
SHOCK (Cardiac disorders) | 0 | 0 | 1
THROMBOSIS (Cardiac disorders) | 0 | 0 | 1
VASCULAR DISORDER (Cardiac disorders) | 1 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 3 | 4 — Digestive System
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 2 | 0
NAUSEA (Gastrointestinal disorders) | 3 | 2 | 2
VOMITING (Gastrointestinal disorders) | 3 | 2 | 1
DIARRHEA (Gastrointestinal disorders) | 1 | 1 | 6
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 | 1 | 0
ILEUS (Gastrointestinal disorders) | 0 | 1 | 1
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0
MUCOSITIS (Gastrointestinal disorders) | 0 | 1 | 2
ANOREXIA (Gastrointestinal disorders) | 1 | 0 | 3
COLITIS (Gastrointestinal disorders) | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 1
GASTROENTERITIS (Gastrointestinal disorders) | 0 | 0 | 1
HEMATEMESIS (Gastrointestinal disorders) | 1 | 0 | 0
HEMORRHAGIC GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 1
HEPATIC FAILURE (Gastrointestinal disorders) | 1 | 0 | 0
HEPATITIS (Gastrointestinal disorders) | 1 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 1
LIVER FATTY DEPOSIT (Gastrointestinal disorders) | 1 | 0 | 0
MELENA (Gastrointestinal disorders) | 1 | 0 | 0
PROCTITIS (Gastrointestinal disorders) | 0 | 0 | 1
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
DIABETES MELLITUS (Endocrine disorders) | 0 | 2 | 0 — Endocrine system
THYROID CARCINOMA (Endocrine disorders) | 1 | 0 | 0
ANEMIA (Blood and lymphatic system disorders) | 12 | 11 | 20 — Hemic and Lymphatic system
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 4
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Blood and lymphatic system disorders) | 0 | 0 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 | 0 | 1
FIBRINOGEN INCREASED (Blood and lymphatic system disorders) | 0 | 0 | 1
THROMBIN TIME PROLONGED (Blood and lymphatic system disorders) | 0 | 0 | 1
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 | 6 | 0 — Metabolic and Nutritional
DEHYDRATION (Metabolism and nutrition disorders) | 7 | 5 | 10
CREATININE INCREASED (Metabolism and nutrition disorders) | 0 | 3 | 1
HYPERCALCEMIA (Metabolism and nutrition disorders) | 2 | 3 | 4
HYPERKALEMIA (Metabolism and nutrition disorders) | 2 | 2 | 2
ALKALINE PHOSPHATASE INCREASED (Metabolism and nutrition disorders) | 0 | 1 | 0
BUN INCREASED (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPERLIPEMIA (Metabolism and nutrition disorders) | 0 | 1 | 3
HYPOCALCEMIA (Metabolism and nutrition disorders) | 0 | 1 | 2
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPONATREMIA (Metabolism and nutrition disorders) | 0 | 1 | 1
PERIPHERAL EDEMA (Metabolism and nutrition disorders) | 1 | 1 | 1
SGOT INCREASED (Metabolism and nutrition disorders) | 0 | 1 | 0
BILIRUBINEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
CACHEXIA (Metabolism and nutrition disorders) | 0 | 0 | 2
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPOGLYCEMIAHYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOPROTEINEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
KETOSIS (Metabolism and nutrition disorders) | 1 | 0 | 0
WEIGHT LOSS (Metabolism and nutrition disorders) | 1 | 0 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 — Musculoskeletal system
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
SPINAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
BONE DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OSTEOPOROSIS FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
CONFUSION (Nervous system disorders) | 3 | 3 | 0 — Nervous system
DIZZINESS (Nervous system disorders) | 0 | 1 | 1
HYPOTONIA (Nervous system disorders) | 0 | 1 | 0
PARESIS (Nervous system disorders) | 0 | 1 | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 1 | 0
AGITATION (Nervous system disorders) | 1 | 0 | 0
AMNESIA (Nervous system disorders) | 1 | 0 | 0
APHASIA (Nervous system disorders) | 0 | 0 | 1
CNS DEPRESSION (Nervous system disorders) | 0 | 0 | 1
CNS NEOPLASIA (Nervous system disorders) | 0 | 0 | 1
COMA (Nervous system disorders) | 1 | 0 | 0
CONVULSION (Nervous system disorders) | 1 | 0 | 1
DELIRIUM (Nervous system disorders) | 1 | 0 | 0
DEPRESSION (Nervous system disorders) | 0 | 0 | 1
DYSTONIA (Nervous system disorders) | 0 | 0 | 1
EXTRAPYRAMIDAL SYNDROME (Nervous system disorders) | 1 | 0 | 0
GRAND MAL CONVULSION (Nervous system disorders) | 1 | 0 | 0
HYPESTHESIA (Nervous system disorders) | 0 | 0 | 1
INSOMNIA (Nervous system disorders) | 1 | 0 | 0
MENTAL STATUS CHANGES (Nervous system disorders) | 0 | 0 | 1
NEUROPATHY (Nervous system disorders) | 1 | 0 | 0
PARALYSIS (Nervous system disorders) | 1 | 0 | 0
PARKINSON'S DISEASE (Nervous system disorders) | 1 | 0 | 0
PSYCHOSIS (Nervous system disorders) | 0 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 1 | 0 | 1
SUICIDAL IDEATION (Nervous system disorders) | 0 | 0 | 1
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 11 — Respiratory system
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 4
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 15
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
CARCINOMA OF LUNG (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
HEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
BRONCHIOLITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
COUGH INCREASED (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
LUNG EDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
LUNG FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
LUNG INFILTRATION NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
SKIN CARCINOMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 — Skin and Appendages
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
CATARACT SPECIFIED (Eye disorders) | 0 | 0 | 2 — Special senses
DIPLOPIA (Eye disorders) | 0 | 0 | 1
ACUTE KIDNEY FAILURE (Renal and urinary disorders) | 6 | 3 | 4 — Urogenital system
GLOMERULITIS (Renal and urinary disorders) | 0 | 1 | 0
KIDNEY FAILURE (Renal and urinary disorders) | 1 | 1 | 3
UREMIA (Renal and urinary disorders) | 0 | 1 | 0
URINARY TRACT INFECTION (Renal and urinary disorders) | 0 | 1 | 0
HEMATURIA (Renal and urinary disorders) | 3 | 0 | 0
KIDNEY FUNCTION ABNORMAL (Renal and urinary disorders) | 1 | 0 | 3
OLIGURIA (Renal and urinary disorders) | 0 | 0 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 2
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 1
URINARY TRACT DISORDER (Renal and urinary disorders) | 1 | 0 | 0
DEVICE MALFUNCTION (General disorders) | 0 | 0 | 2 — Adverse event associated with miscellaneous factors
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Alfa (N=200) | Temsirolimus (N=208) | Interferon Alfa and Temsirolimus (N=208)
ASTHENIA (General disorders) | 126 | 105 | 127 — Body as a whole
PAIN (General disorders) | 30 | 56 | 41
FEVER (General disorders) | 98 | 49 | 126
ABDOMINAL PAIN (General disorders) | 34 | 42 | 34
BACK PAIN (General disorders) | 28 | 41 | 31
CHEST PAIN (General disorders) | 18 | 35 | 23
HEADACHE (General disorders) | 30 | 32 | 47
INFECTION (General disorders) | 11 | 29 | 32
ALLERGIC REACTION (General disorders) | 1 | 18 | 11
CHILLS (General disorders) | 58 | 17 | 72
FACE EDEMA (General disorders) | 1 | 15 | 10
ACCIDENTAL INJURY (General disorders) | 8 | 13 | 12
FLU SYNDROME (General disorders) | 23 | 8 | 28
LAB TEST ABNORMAL (General disorders) | 5 | 8 | 13
HYPERTENSION (Cardiac disorders) | 7 | 12 | 12 — Cardiovascular system
HYPOTENSION (Cardiac disorders) | 11 | 10 | 7
TACHYCARDIA (Cardiac disorders) | 11 | 9 | 17
VASODILATATION (Cardiac disorders) | 5 | 5 | 12
NAUSEA (Gastrointestinal disorders) | 82 | 76 | 84 — Digestive system
ANOREXIA (Gastrointestinal disorders) | 86 | 66 | 79
DIARRHEA (Gastrointestinal disorders) | 39 | 57 | 56
CONSTIPATION (Gastrointestinal disorders) | 35 | 42 | 39
STOMATITIS (Gastrointestinal disorders) | 7 | 41 | 42
MUCOSITIS (Gastrointestinal disorders) | 10 | 39 | 46
VOMITING (Gastrointestinal disorders) | 57 | 39 | 60
DRY MOUTH (Gastrointestinal disorders) | 16 | 13 | 12
MOUTH ULCERATION (Gastrointestinal disorders) | 5 | 6 | 15
ORAL MONILIASIS (Gastrointestinal disorders) | 4 | 5 | 15
ANEMIA (Blood and lymphatic system disorders) | 78 | 90 | 123 — Hemic and Lymphatic system
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 16 | 28 | 77
NEUTROPENIA (Blood and lymphatic system disorders) | 26 | 15 | 57
LEUKOPENIA (Blood and lymphatic system disorders) | 34 | 13 | 65
LYMPHOPENIA (Blood and lymphatic system disorders) | 17 | 11 | 28
HYPERLIPEMIA (Metabolism and nutrition disorders) | 29 | 57 | 80 — Metabolic and Nutritional
PERIPHERAL EDEMA (Metabolism and nutrition disorders) | 15 | 54 | 36
HYPERCHOLESTEREMIA (Metabolism and nutrition disorders) | 9 | 51 | 55
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 22 | 49 | 36
WEIGHT LOSS (Metabolism and nutrition disorders) | 49 | 40 | 65
CREATININE INCREASED (Metabolism and nutrition disorders) | 21 | 28 | 42
ALKALINE PHOSPHATASE INCREASED (Metabolism and nutrition disorders) | 15 | 20 | 31
HYPOKALEMIA (Metabolism and nutrition disorders) | 7 | 20 | 14
EDEMA (Metabolism and nutrition disorders) | 8 | 19 | 8
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 4 | 17 | 21
SGOT INCREASED (Metabolism and nutrition disorders) | 29 | 16 | 43
HYPOPROTEINEMIA (Metabolism and nutrition disorders) | 18 | 13 | 21
LACTIC DEHYDROGENASE INCREASED (Metabolism and nutrition disorders) | 7 | 12 | 19
SGPT INCREASED (Metabolism and nutrition disorders) | 14 | 12 | 15
HYPOCALCEMIA (Metabolism and nutrition disorders) | 21 | 11 | 32
HYPERCALCEMIA (Metabolism and nutrition disorders) | 11 | 8 | 8
HYPERKALEMIA (Metabolism and nutrition disorders) | 18 | 8 | 11
DEHYDRATION (Metabolism and nutrition disorders) | 15 | 7 | 22
HYPONATREMIA (Metabolism and nutrition disorders) | 7 | 6 | 15
BUN INCREASED (Metabolism and nutrition disorders) | 5 | 3 | 11
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 29 | 38 | 27 — Musculoskeletal system
MYALGIA (Musculoskeletal and connective tissue disorders) | 30 | 16 | 22
BONE PAIN (Musculoskeletal and connective tissue disorders) | 11 | 8 | 7
INSOMNIA (Nervous system disorders) | 29 | 25 | 36 — Nervous system
DIZZINESS (Nervous system disorders) | 25 | 18 | 27
ANXIETY (Nervous system disorders) | 12 | 16 | 24
PARESTHESIA (Nervous system disorders) | 10 | 14 | 13
SOMNOLENCE (Nervous system disorders) | 21 | 14 | 14
DEPRESSION (Nervous system disorders) | 26 | 9 | 25
CONFUSION (Nervous system disorders) | 17 | 6 | 10
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 42 | 59 | 51 — Respiratory system
COUGH INCREASED (Respiratory, thoracic and mediastinal disorders) | 29 | 55 | 49
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 7 | 27 | 27
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 3 | 24 | 27
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 4 | 20 | 10
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 1 | 14 | 7
RASH (Skin and subcutaneous tissue disorders) | 11 | 76 | 34 — Skin and Appendages
PRURITUS (Skin and subcutaneous tissue disorders) | 16 | 40 | 24
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 | 28 | 5
DRY SKIN (Skin and subcutaneous tissue disorders) | 14 | 22 | 13
ACNE (Skin and subcutaneous tissue disorders) | 2 | 21 | 7
EXFOLIATIVE DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 16 | 6
PRURITIC RASH (Skin and subcutaneous tissue disorders) | 1 | 11 | 3
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 1 | 11 | 6
SWEATING (Skin and subcutaneous tissue disorders) | 14 | 5 | 15
TASTE PERVERSION (General disorders) | 13 | 31 | 18 — Special Senses
TASTE LOSS (General disorders) | 4 | 11 | 5 — Special Senses
URINARY TRACT INFECTION (Renal and urinary disorders) | 10 | 16 | 23 — Urogenital system

LIMITATIONS AND CAVEATS:
Efficacy data was not collected or analyzed after the primary analysis was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.